CLINICAL TRIAL: NCT06931808
Title: The Efficacy and Safety of Intestinal Microbiota Transplantation Combined With Radiochemotherapy and Sintilimab in Neoadjuvant Treatment for Locally Advanced Rectal cancer-a Single Arm, Prospective, Single Center Exploratory Study
Brief Title: Intestinal Microbiota Transplantation, Radiochemotherapy and Sintilimab in Localized Advanced Colon Cancer
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Qingsong Tao, chief physician, First Affiliated Hospital of Ningbo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-XM-038
Record Dates: First submitted 2025-03-15; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Localized Advanced Rectal Adenocarcinoma
Keywords: mid-low position; IIA-IIIC (T3-4/N+)
MeSH Terms: interventions — sintilimab; Drug Therapy; Gastrointestinal Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intestinal microbiota transplantation combined with chemoradiotherapy and Sintilimab (Experimental): Intestinal microbiota transplantation combined with synchronous radiotherapy, chemotherapy, and Sintilimab as neoadjuvant therapy
  Interventions: Drug: Sintilimab plus Chemotherapy; Drug: Intestinal microbiota capsules; Radiation: Standard Long Course Radiotherapy; Procedure: Total mesorectal excision

INTERVENTIONS:
Drug: Sintilimab plus Chemotherapy — All patients received standard long-term radiation therapy (LCRT) (50.0Gy/25f) and concurrent chemotherapy with capecitabine (825 mg/m2, bid, po) (Phase 1); Xelox scheme (Oxaliplatin 130 mg/m2, ivgtt ，d1； Capecitabine 1000 mg/m2, bid，d1-14) (Phase 2); . During the radiotherapy and chemotherapy period, they also received two cycles of immunotherapy with Sintilimab (200mg, ivgtt, d1, q3w).
Drug: Intestinal microbiota capsules — During Phase 1, intestinal microbiota transplantation treatment, oral intestinal microbiota capsules are used for transplantation treatment, with a dose of 30 capsules/day (about 1U sediment microbiota, containing about 1 × 1013 bacteria). Transplantation is carried out continuously for 3 days starting from each week, for a total of 3 courses of treatment.
Radiation: Standard Long Course Radiotherapy — 50.0Gy/25f
Procedure: Total mesorectal excision — 6-8 weeks after the end of the first phase and combined with 5 cycles of Xelox regimen adjuvant chemotherapy.

SUMMARY:
The standard treatment for locally advanced rectal cancer is neoadjuvant chemoradiotherapy followed by total mesorectal excision. While Immune checkpoint inhibitors are promising in the treatment of various cancers, the combination of radiotherapy and immunotherapy still lacks high-level evidence-based medicine, and the efficacy is still limited in rectal cancer.

Thus, we designed a study on the efficacy and safety of intestinal microbiota transplantation combined with synchronous radiochemotherapy and immune checkpoint inhibitor xindilimab neoadjuvant therapy for locally advanced rectal cancer.

DETAILED DESCRIPTION:
The incidence rate of colorectal cancer (CRC) ranks among the top three most common cancers in the world, while the mortality rate ranks among the top two. Early symptoms of rectal cancer are not obvious, and about 60% of patients are diagnosed with locally advanced rectal cancer. The standard treatment for locally advanced rectal cancer is neoadjuvant chemoradiotherapy followed by total mesorectal excision. However, the response of patients to radiotherapy showed significant heterogeneity, with pathological complete response rates (pCR) ranging from 6% to 39%. In addition, a significant proportion of LARC patients (20% -40%) do not respond to preoperative radiotherapy (preRT). Therefore, it is crucial to find ways to alleviate radiation resistance within tumors.

Immune checkpoint inhibitors (ICIs) are increasingly being used in various solid tumors. However, immunotherapy in the field of CRC has always been distinct, with patients with mismatch repair defects (dMMR) or high microsatellite instability (MSI-H) (accounting for 5% -15% of all CRCs) having a higher tumor mutation burden (TMB) and more tumor infiltrating lymphocytes (TILs), making them the absolute dominant population for immunotherapy; However, patients with microsatellite stability (MSS) or normal mismatch repair (pMMR) have poor immune therapy efficacy. At present, radiotherapy is widely regarded as a mechanism that triggers local and systemic immune responses, providing a theoretical basis for the combination of radiotherapy and immunotherapy (iRT). In 2022, the VOLTAGE-A study reported the addition of nivolumab treatment after long-term synchronous chemoradiotherapy. The results showed that the major pathological response (MPR) rate and pCR rate in 37 MSS LARC patients after surgery were 38% and 30%, respectively. In addition, multiple studies have conducted similar explorations with different methods. Overall, these studies have achieved certain therapeutic effects, with pCR rates ranging from 37.5% to 57.1%. However, the combination of radiotherapy and immunotherapy still lacks high-level evidence-based medicine, and the efficacy is still limited.

The gut microbiota is a complex microbial community closely related to the occurrence and development of rectal cancer. Previous studies have shown that gut microbiota can predict response to neoadjuvant radiotherapy, improve treatment response, and reduce treatment toxicity. In addition, it has been confirmed that the gut microbiota can reshape the tumor immune microenvironment (TiME), thereby affecting the response to ICIs. The results of two Phase I trials indicate that gut microbiota transplantation (FMT) derived from responders effectively reversed immune resistance in melanoma, laying the foundation for the clinical application of FMT in cancer immunotherapy. In a phase II study, a total of 20 MSS mCRC patients were enrolled and received FMT combined with trastuzumab and furosemide as third line or above treatment. The median PFS was 9.6 months (95% CI 4.1-15.1) and the median OS was 13.7 months (95% CI 9.3-17.7), with controllable side effects, demonstrating the potential of FMT in the field of rectal cancer.

ELIGIBILITY:
1. Must sign the informed consent form with good compliance;
2. Age 18 to 75 years ;
3. ECOG score 0-1 points;
4. Locally advanced rectal adenocarcinoma and TNM clinical stage IIA-IIIC (T3-4/N+);
5. The distance between the lower edge of the tumor and the anal margin is less than or equal to 10cm.
6. Have not received any anti-tumor treatment in the past (including but not limited to surgery, radiotherapy, chemotherapy, anti vascular therapy, immunotherapy, etc.); 7 The main organ functions well. -

Exclusion Criteria:

* 1. Other malignant tumors, including rectal cancer with other pathological types within 5 years; 2. Not using probiotics in the past 2 months; 3. Severe damage to the intestinal barrier, such as sepsis, active gastrointestinal bleeding, perforation, etc.; 4. Weight loss of ≥ 20% within 90 days; 5. Poor nutritional status or PG-SGA score ≥ 9; 6. Severe and/or uncontrolled illnesses.

  1. Poor blood pressure control (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 100mmHg)
  2. ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (QTc ≥ 470ms), and ≥ grade 2 congestive heart failure
  3. History of interstitial lung disease, non infectious pneumonia, pulmonary fibrosis, or other uncontrolled acute lung diseases
  4. Active or uncontrolled severe infection (≥ CTCAE level 2 infection)
  5. Cirrhosis and active hepatitis; Active hepatitis (hepatitis B reference: HBsAg is positive, and the HBV DNA detection value exceeds the upper limit of normal value; Hepatitis C reference: HCV antibody positive and HCV virus titer detection value exceeding the upper limit of normal); Note: Subjects with positive hepatitis B B surface antigen or core antibody and patients with hepatitis C who meet the inclusion conditions need continuous antiviral treatment to prevent virus activation
  6. Active syphilis patients
  7. Renal failure requiring hemodialysis or peritoneal dialysis
  8. History of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases, or organ transplantation 7. Poor control of diabetes (fasting blood glucose [FBG]>10mmol/L) 8. Significant surgical treatment, open biopsy, or significant traumatic injury within 60 days prior to the start of treatment; Or long-term untreated wounds or fractures 9. Serious arterial/venous thrombotic events such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism occurred within 6 months before the start of treatment 10. History of abuse of psychotropic drugs who are unable to quit or have mental disorders 11. History of severe allergies 12. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response rate | Up to 12 weeks
  Defined as the percentage of subjects with ypT0N0 who have no residual tumor cells in the primary tumor and lymph nodes after surgery compared to all subjects.
Overall Survival | Three years after the end of treatment
  The percentage of subjects who are still alive after 3 years of follow-up among all subjects.
R0 resection rate | During the surgery
  Defined as the complete resection rate of tumors with negative margins removed under a microscope
Tumor regression grading | During the surgery
  According to AJCC 8th edition, the Tumor regression grading is based on the proportion of fibrosis and residual tumors in the tumor. Grade 0 indicates complete regression of the tumor, Grade 1 indicates regression of over 90%, Grade 2 indicates regression between 10% and 90%, Grade 3 indicates regression of less than 10%, and Grade 4 indicates no significant regression of the tumor
Completion rate of neoadjuvant therapy | Up to 6 weeks
  Defined as the percentage of subjects who have completed all neoadjuvant therapies compared to all subjects
Event free survival rate | Three years after the end of treatment
  The percentage of subjects who were followed up for 3 years and still survived without disease recurrence or change of treatment plan among all subjects.
Disease-free survival rate | Three years after the end of treatment
  The percentage of subjects who were followed up for 3 years and still survived without disease recurrence among all subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China